CLINICAL TRIAL: NCT06405737
Title: Oxytocin Modulates the Processing of the Advantageous- and Disadvantageous-inequity
Brief Title: Oxytocin's Effect on the Advantageous- and Disadvantageous-inequity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Shuxia Yao, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-88
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: advantageous inequity; disadvantageous inequity; fMRI; oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin (Experimental): a single dose of 24 international units (IU) of OT will be administered with 3 puffs of treatment to each nostril.
  Interventions: Drug: Intranasal oxytocin
- placebo (Experimental): a single dose of 24 international units (IU) of placebo will be administered with 3 puffs of treatment to each nostril.
  Interventions: Drug: Intranasal placebo

INTERVENTIONS:
Drug: Intranasal oxytocin — Subject assigned to receive intranasal administration of oxytocin (24 IU).
  Arms: oxytocin
Drug: Intranasal placebo — Subjects assigned to receive intranasal administration of placebo (24 IU).
  Arms: placebo

SUMMARY:
The main aim of the study is to investigate whether intranasal oxytocin modulates advantageous- and disadvantageous-inequity and whether oxytocin has similar effects on them or not.

DETAILED DESCRIPTION:
The main aim of the study is to investigate whether intranasal oxytocin modulates advantageous- and disadvantageous-inequity and its underlying neural mechanisms and whether oxytocin has similar effects on them or not. A double-blinded, placebo-controled, between-subject design is employed in this study. In a randomized order, a total of 80 healthy males are instructed to self-administrated intranasal spray of oxytocin or placebo. A modified inequity decision-making task starts 45 minutes after treatment with behavioral (fairness rating, preference rating and the choice rate of unequal option) and fMRI data being collected during this task. Personality traits of subjects are assessed using validated Chinese version questionnaires including the Beck Depression Inventory (BDI-II), State-Trait Anxiety Inventory (STAI), Autism Spectrum Quotient (ASQ), Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ), Behavioral Inhibition System and Behavioral Activation System Scale (BIS/BAS). Subjects are asked to complete Positive and Negative Affect Schedule (PANAS) when they just arrive, before and after the task.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury
* pregnant,menstruating,taking oral contraceptives
* medical or psychiatric illness.
* excessive head movement (> 3mm) during scanning

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Behavioral index: fairness rating scores | 45-75 minutes after treatment administration
  Participants are instructed to rate their perceived levels of fairness to the allocation using a 9-point Likert scale within 4 seconds (1 = very unfair, 9 = very fair).
Behavioral index: preference rating scores | 45-75 minutes after treatment administration
  Participants are instructed to rate their perceived levels of preference to the allocation using a 9-point Likert scale within 4 seconds (1 = not at all, 9 = very preferable).
Neural indices: fMRI-based measures of the outcome presentation stage | 45-75 minutes after treatment administration
  Functional magnetic resonance imaging (fMRI) is employed to assess participants' blood-oxygen-level dependent signals when they are confronted with monetary allocations (advantageous-inequity, disadvantageous-inequity, and fair).

SECONDARY OUTCOMES:
Behavioral index: choice rate of unequal option | 45-75 minutes after treatment administration
  Participants are instructed to make a hypothetical choice between the actual allocation in the current trial and the other fair option if they were given another chance to re-choose.
Neural indices: fMRI-based measures of outcome and re-decision stages | 45-75 minutes after treatment administration
  Functional magnetic resonance imaging (fMRI) is employed to assess participants' blood-oxygen-level dependent signals when they are instructed to make a hypothetical choice between the actual allocation in the current trial and the other fair option if they were given another chance to re-choose.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Shuxia, Dr, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China (UESTC), Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No